CLINICAL TRIAL: NCT01337895
Title: Diet and Weight Loss Study - a Weight Loss Trial to Determine Whether Dairy Products Augment Weight Loss for Adults Following an Energy-restricted Weight Loss Study
Brief Title: DAWL (Dairy and Weight Loss) Study
Acronym: DAWL
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Grant not funded, study will not launch
Sponsor: University of Guelph (Other)
Collaborators: Purdue University (Other); University of Saskatchewan (Other)
Responsible Party: Andrea Buchholz, University of Guelph
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11MR010
Record Dates: First submitted 2011-04-15; First posted 2011-04-19 (Estimated); Last update posted 2011-11-11 (Estimated); Status verified 2011-08

CONDITIONS: Obesity; Overweight
Keywords: Dairy; obesity; overweight; weight loss; adults
MeSH Terms: conditions — Obesity; Overweight; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lifestyle counselling (Active Comparator): These participants will be assigned to a 500 kcal/day energy-restricted diet that is low in dairy products (no more than 1 serving per day).
  Interventions: Other: Low dairy
- High dairy (Experimental): These participants will be assigned a 500 kcal/day energy-restricted diet that is high in dairy (4 or more servings per day).
  Interventions: Other: High dairy

INTERVENTIONS:
Other: Low dairy — No more than 1 serving per day
  Arms: Lifestyle counselling
Other: High dairy — 4 or more servings per day
  Arms: High dairy

SUMMARY:
* Objectives Taking a 'whole foods' approach, we will investigate (i) whether consumption of isocaloric diets containing ≥4 vs. ≤1 servings of dairy products per day for 16 weeks results in greater body fat loss in energy-restricted overweight/obese premenopausal women; (ii) the role of dairy product consumption in influencing physiological and metabolic factors which may precede or accompany changes in body composition, including in enzymes which synthesize and break down body fat; and (iii) factors, including obesity phenotype, which may influence the response of body composition to dairy product consumption.
* Background

With the obesity epidemic showing no signs of abating, there is ongoing interest, both at the lay public and scientific levels, in manipulating the diet to promote weight, specifically fat, loss. One such promising manipulation is an increase in, or perhaps more precisely, an isocaloric substitution of, dairy product consumption. The inverse association between Body Mass Index (BMI) and dietary calcium - for which dairy products are the main source - was first described in 1984 and has since been supported by various levels of evidence, but not consistently. Heaney recently described this literature as "confused," which he and Rafferty attribute to important limitations in study design, including lack of low-calcium contrast groups and the fact that body weight/body composition is often a secondary endpoint in studies designed and powered for a different outcome, typically bone health or blood pressure. Confusion has also arisen from the investigation of different interventions (dairy products, dairy calcium, dietary calcium, supplemental calcium), making it difficult to compare and interpret studies. This creates an opportunity for the proposed Dairy and Weight Loss (DAWL) study, with its focus on whole dairy product consumption, to help clear up the confusion surrounding this issue.

**Hypotheses

Overweight/obese, low habitual dairy consuming, premenopausal women randomized to an energy-restricted weight loss diet containing ≥4 servings/day of dairy products (milk, yogurt, cheese) for 16 weeks will lose more body fat than those randomized to an isocaloric diet containing ≤1 servings/day of dairy products.

DETAILED DESCRIPTION:
"Ground zero" for the DAWL study will be the University of Guelph Body Composition and Metabolism Lab (www.uoguelph.ca/bodycomp), under the direction of the PI.

Sample Size. The investigators plan to complete data collection on a total of 46 women. This sample size is based on an anticipated total body fat mass (FM) loss over 16 weeks of 5.5 kg in the high dairy group and 3.8 kg in the control group. These values are based on data published from 4 studies (5; 20-22). To be conservative in our sample size calculation, we used a higher-than-reported SD of 2.0 kg FM loss. Together, these values indicated that we require 23 women in each group to detect a significant difference in total body FM, with 80% power and 5% alpha. Attrition and non-adherence is anticipated to be approximately 20% to 25%, therefore 30 women in each group will be recruited. We anticipate screening approximately 300+ women to collect 16 weeks of data on a total of 46 eligible and adherent completers, as per Figure 1 below.

Inclusion/Exclusion Criteria. Inclusion criteria include non-smoking, non-pregnant and non-lactating women 18 to 50 years; premenopausal (determined by cessation of menstruation and recent menstrual history to exclude those who are perimenopausal or amennorheic); BMI ≥25.0 kg/m2 (54); usual calcium consumption below the EAR of 800 mg/d (55) to be measured using a validated calcium and vitamin D food frequency questionnaire (FFQ) (56); no sensitivity to dairy; normal liver and kidney function, serum calcium, and complete blood count; 3 mo history of weight stability; and willingness to adhere to study protocol for 16 weeks regardless of treatment, and including no change in physical activity levels. Any vitamin/mineral supplement users will be asked to discontinue supplementation for 4 weeks prior to enrolling in the trial (i.e. "wash out"), as well as for the duration of the trial.

Exclusion criteria include violation of any of the above, or presence of a health condition which might influence weight loss (such as diabetes, CVD, cancer, thyroid disease) or regularly taking medication which may do the same (such as corticosteroids).

Comprehensive Screening/Background Data Collection Visit. Women who pass the initial screen and attend the recruitment session will be invited back to the lab, after having fasted for 12 hours (no food or drink except water), where they will first be asked to sign an informed consent form. Further screening/background data to be collected will include:

* Biochemistry including complete blood count, liver function tests (ALT, AST), blood urea nitrogen, creatinine, and serum total calcium. Participants will undergo venipuncture by a LifeLabs phlebotomist (letter of support attached). A 3 business day turnaround is anticipated for results. Participants with values within normal limits will continue on to enrollment. By this stage of recruitment, participants with any known health conditions/medications suspected to interfere with study outcomes will have been screened out, therefore it is anticipated that most will have values within normal limits.
* International Physical Activity Questionnaire (IPAQ) (57) to assess usual activity habits.
* Resting metabolic rate (kcal/d) to determine the energy levels of individualized meal plans, which will be calculated as (RMR x PAL) - 500 kcal/d. RMR will be measured using continuous open-circuit indirect calorimetry using a MAX-IIa instrument (AEI Technologies Inc.). RMR measurements will be conducted with participants lying awake but at complete physical rest, with a ventilated hood placed over the head and neck. Participants will undergo measurement for 30 to 40 minutes; the first 5 to 10 minutes of data will be discarded to allow for acclimation to the testing environment. We will provide a juice box and granola bar after this test so that participants are not hungry. For consistency across study visits, we will measure participants in the follicular phase of their menstrual cycles.

14.5 Lead-In Phase During the two weeks following the comprehensive screening visit, participants will be asked maintain a 3-day food record, from which research personnel will create 500 kcal-restricted individualized meal plans as described below. From this point on, participants will be asked to maintain their usual physical activity levels.

14.6 Study Diets Participants will be provided with individualized meal plans - high dairy or control - every two weeks for the duration of the study. They will be counseled on their assigned diets by research personnel during the baseline visit and throughout the study. The energy levels of the meal plans (e.g. 1200 kcal, 1400 kcal, 1600 kcal, etc) will be determined from RMR and PAL levels as follows: (RMR x PAL) - 500 kcal/d, where RMR is resting metabolic rate (kcal/d, measured by indirect calorimetry), PAL is physical activity level derived from the screening IPAQ and 500 kcal is the daily energy restriction. The energy levels will be adjusted throughout the study as needed. Actual foods in the meal plans will be based on Eating Well with Canada's Food Guide (EWCFG, http://www.hc-sc.gc.ca/fn-an/food-guide-aliment/index-eng.php) and the 3-day food records completed during the lead-in phase. The diets for the two treatment groups will be matched for energy and macronutrient (protein, fat, carbohydrate) intake as per the sample 1400 kcal meal plans attached, and using ESHA Food Processor SQL (version 10.8.0, ESHA Research, Salem OR) updated with the 2010 Canadian Nutrient File.

Dairy products for the high dairy group will be donated by Agropur Coopérative and Ultima Foods (letter of support attached). Consistent with EWCFG recommendations, a variety of dairy products (milk, yogurt, cheese) will be included. One serving will be considered 1 cup fluid white cow's milk or chocolate milk; 1.5 ounces cheese; and 1 cup yogurt. Although EWCFG considers 1 serving of yogurt to be 0.75 cups, we will increase to 1 cup to provide equivalent calcium across all dairy products. Minimum dairy calcium intake of the high-dairy group is anticipated to be 1200 mg/d; dietary calcium intake will be higher. Dietary calcium of the control group is anticipated to be <450 mg/d, therefore we anticipate a spread of approximately 1000 mg dietary calcium per day between groups. If energy levels of meal plans allow, we will incorporate regular fat (vs. low fat) dairy products to reflect Canadians' actual dairy intake and maximize intake of CLA. Participants in the high-dairy group will be provided with a 2 week supply of dairy products at a time, in insulated transport bags.

14.7 Baseline Visit (week 0)

Following lead-in, participants will return to the lab for a baseline visit. At this time, participants will first be informed to which treatment they were randomly assigned by the biostatistician (using a random number generator) and to which they will be asked to adhere for 16 weeks. We will divulge this prior to going any further, to provide an opportunity for participants to withdraw. Willing participants will then undergo a series of measurements:

* Weight as described above.
* Waist circumference will be measured twice on standing participants at the level of the iliac crest (58) using a Gulick II non-elastic tape measure; if measures differ by > 5%, a third will be taken and the mean of the two closest values will be used. Hip circumference will be measured twice on standing participants around the widest portion of the buttocks (59); if measures differ by >5%, a third will be taken and the mean of the two closest values will be used. Predominantly android obesity will be defined as a waist-to-hip ratio of >0.85, predominantly gynoid obesity will be defined as a waist-to-hip ratio of ≤0.85 (59, 60).
* Body composition. Whole body and regional fat mass and lean mass will be measured by dual energy x-ray absorptiometry (DXA) using a fan beam Hologic Wi updated with APEX 3.2 software. See Figure 2. Participants will be asked to wear underpants and a hospital gown only, and to remove all metal jewelry, for this test
* Venipuncture. A LifeLabs phlebotomist will draw fasting blood samples from each participant. Biochemical analyses to be completed at LifeLabs include glucose, insulin, 25(OH)D, lipids (total cholesterol; HDL; LDL; triglycerides), high-sensitivity C-reactive protein (hsCRP), and parathyroid hormone (PTH). Various CLA isomers (c9, t11; t10, c12) in red blood cells (Dr. David Ma), and hepatic lipase, lipoprotein lipase and mRNA expression of fatty acid synthase (Dr. Marica Bakovic) will be analyzed in yearly batches at the University of Guelph. Participants are required to fast for this visit; we will provide a juice box and granola bar afterwards.
* Visual analog scale (VAS) to assess desire to eat, hunger, fullness and prospective food consumption (61). Scales are 100 mm in length and are anchored at either end with words expressing the most positive and negative ratings. The VAS will be completed in the lab conference room after venipuncture.
* Sitting blood pressure using a digital blood pressure cuff (Physio Logic model 106-94, Montréal PQ).

14.8 Mid-Study Visit (week 8) Participants will repeat the following tests: weight, waist/hip circumferences, DXA, resting metabolic rate, blood pressure.

14.9 Study Conclusion (week 16) Participants will repeat all of the same tests as during the Baseline Visit. 14.10 Adherence and Interim Visits Throughout the trial, participants will maintain a daily dairy product intake checklist and weekly food and activity diaries to determine adherence to treatment group, energy intake and physical activity. Biweekly, participants will visit the lab to turn in checklists; have meal plans reassessed; and have weight, BMI and waist/hip circumferences measured. Those in the dairy group will pick up a 2 week supply of dairy products. Participants will complete a monthly calcium and vitamin D FFQ (56).

14.11 Data Analysis Repeated measures ANOVA will be conducted for all measures collected at more than two time points, to determine differences between treatment groups. These include: body composition (DXA, weight, BMI, waist/hip circumferences), dietary data, physical activity, resting metabolic rate, visual analog scale and blood pressure. Consistent with a pre/post design, paired t-tests will determine differences in biochemical variables measured at weeks 0 and 16. Regression analyses will be used to predict kilograms of fat mass lost, with predictor variables including obesity phenotype (predominantly android vs. predominantly gynoid adjusted for any differences in BMI), baseline 25(OH)D status, age, etc.

14.12 Knowledge Translation

Community, provincial and national outreach to consumers, Registered Dietitians (RD), other health care professionals, and scientists will be achieved through multiple means:

* Gwen Laughton and Janine Robertson, Guelph-based RD collaborators, will provide KT assistance specifically tailored to the local context. This includes presentations and discussion groups with other Guelph-based RDs to assist with health literacy for consumers, and dissemination via the Waterloo Wellington Regional Nutrition Network. We will also post the study on the web-based Ontario Nutrition Resource Centre, an initiative of the Ontario Public Health Association.
* The DAWL study will be posted on the Canadian Inventory of Nutrition and Dietetic Associated Research (CINDAR) and Canadian Obesity Network (CON) websites, and in the "Members in Action" section of the Dietitians of Canada newsletter. The PI, co-investigators and graduate students will collaborate on scientific publications and presentations at nutrition meetings (e.g. Canadian Nutrition Society). The research team will work with media specialists to reach and educate the public, and with the agri-food chain (industry, not-for-profit trade association, marketing group) including Dairy Farmers of Canada, Agropur Coopérative and Ultima Foods, Dairy Farmers of Ontario, Ontario Dairy Council.

ELIGIBILITY:
Inclusion Criteria:

* Otherwise healthy adult premenopausal women with a Body Mass Index (BMI) equal to or greater than 25 kg/m2
* Age 18 to 50 years
* Healthy, to be determined from a background health questionnaire and a screening blood panel
* Willing to comply with study protocol
* able to visit laboratory regularly throughout the study (therefore must live within reasonable driving distance of the University of Guelph)

Exclusion Criteria:

* Presence of any disease which may interfere with study outcomes including cardiovascular disease, diabetes, cancer, thyroid problem, renal disease, liver disease
* not be willing to comply with study protocol

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2012-05; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Body fat | 16 weeks
  Whole body fat will be measured at baseline (Week 0) and follow-up (Week 16) by dual energy x-ray absorptiometry

SECONDARY OUTCOMES:
Body weight | 16 weeks
  The investigators will measure body weight every 2 weeks during the trial
Body mass index (BMI) | 16 weeks
  Body mass is weight (in kg) divided by height (in m2), to be measured every 2 weeks
Waist and hip circumference | 16 weeks
  The investigators will measure waist and hip circumference, using a measuring tape, every 2 weeks throughout the trial.
Fat-free mass | 16 weeks
  Similar to fat mass, the investigators will measure fat-free mass at weeks 0 and 16, using dual energy x-ray absorptiometry
Biochemistry | 16 weeks
  The investigators will measure various biochemical variables at weeks 0 and 16. These will include: glucose, insulin, lipid panel (triglyeride, total cholesterol, HDL cholesterol, LDL cholesterol), vitamin D, parathyroid hormone, C-reactive protein, conjugated linoleic acid concentrations of red blood cells, and hepatic lipase and lipoprotein lipase
Blood pressure | 16 weeks
  The investigators will measure blood pressure every two weeks during the study.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea C. Buchholz, PhD, RD, Principal Investigator — University of Guelph
Locations (1):
- Body Composition and Metabolism Lab, University of Guelph, Guelph, Ontario, Canada